CLINICAL TRIAL: NCT05786235
Title: Patients Pregnant Women With or Without Primary Antiphospholipid Antibody Syndrome
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, Associate Professor of Internal Medicine, Vita-Salute San Raffaele University Head physician, U.O. General Medicine and Continuity of Care, IRCCS San Raffaele Hospital, IRCCS San Raffaele
Other Study IDs: APS_FLT1/PLGF
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Preeclampsia; Immunologic Disease; Antiphospholipid Antibody Syndrome Primary; Pregnancy Complications; Pregnancy, High Risk; Rheumatic Diseases
MeSH Terms: conditions — Pre-Eclampsia; Immune System Diseases; Pregnancy Complications; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant patients with primary APS: Diagnosis of primary APS, according to international classification criteria
  Interventions: Other: Collection of epidemiological and anamnestic data and collection of biological material (peripheral blood)
- pregnant patients who do not have APS: Patients with at least one previous full-term pregnancy No diagnosis of APS, according to international classification criteria
  Interventions: Other: Collection of epidemiological and anamnestic data and collection of biological material (peripheral blood)

INTERVENTIONS:
Other: Collection of epidemiological and anamnestic data and collection of biological material (peripheral blood) — Patients will be enrolled in the study during the first trimester of gestation or later, if the diagnosis of APS is made during pregnancy followed by clinical practice. During the quarterly visits scheduled by clinical practice, the following will be collected relevant clinical information and the additional biological samples for analysis of serum levels of sFlt-1 and PlGF. A follow-up postpartum visit is scheduled by clinical practice at 6 weeks after completion of delivery.
  Groups: pregnant patients with primary APS
Other: Collection of epidemiological and anamnestic data and collection of biological material (peripheral blood) — Patients will be enrolled during the performance of prenatal diagnosis, routinely chosen by the patient, at which the relevant clinical information and the additional biological sample . Collection of biological material in the 2nd and 3rd TM of gestation will take place at occasion of the routinely scheduled ultrasound scans . A postpartum follow-up visit is scheduled by clinical practice at 6 weeks after the completion of delivery.
  Groups: pregnant patients who do not have APS

SUMMARY:
The purpose of the study is to evaluate the ability of placental angiogenesis markers to predict the risk of PE in pregnancy in women with primary APS.

To construct reference intervals of placental angiogenesis markers specific to women affected by primary APS in pregnancy by measuring the levels of sFlt-1and PlGF in serum maternal serum and their sFlt-1/PlGF ratio during the trimesters of gestation (I TM, II TM and III TM).

For this aim the study will involve recruiting two groups of subjects, one will be cases and one will be controls.

ELIGIBILITY:
Inclusion Criteria:

* Group 1

  1. Pregnant patients between the ages of 18 and 45 years.
  2. Diagnosis of primary APS, according to international classification criteria.
* Group 2

  1. Pregnant patients between the ages of 18 and 45 years.
  2. Patients with at least one previous full-term pregnancy.
  3. No diagnosis of APS, according to international classification criteria.

Exclusion Criteria:

* Group 1

  1. PMA pregnancies.
  2. Known chronic pathology in gestational period such as chronic essential hypertension, neurological pathology
  3. Previous thrombotic event
  4. Chronic renal failure not related to AD
  5. Previous history of oncology
* Group 2

  1. Pregnancy by PMA.
  2. Previous history of polyabortion and/or late pregnancy complications.
  3. Known chronic pathology in gestational period such as chronic essential hypertension, neurological pathology
  4. Previous thrombotic event
  5. Previous history of oncology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: At least 60 patients aged 18-45 years will be enrolled between the first and third trimester of gestation, specifically 40 pregnant patients with primary APS (Group 1) and 20 pregnant patients without APS (Group 2) followed at the outpatient clinics of Obstetrics and Pregnancy Pathology of the participating centers. All patients will be asked to sign an informed consent prior to the collection of data and biological material.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
To construct reference ranges of placental angiogenesis markers specific to women with primary APS in pregnancy | six month after the end of the study
  To construct reference ranges of placental angiogenesis markers specific to women with primary APS in pregnancy by measuring the levels of sFlt-1and PlGF in serum maternal serum and their sFlt-1/PlGF ratio during the trimesters of gestation (I TM, II TM and III TM).

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided